CLINICAL TRIAL: NCT03239808
Title: Assessment of the Incremental Haemodialysis Security and Effectiveness in Incident Patients
Brief Title: Incremental Haemodialysis in Incident Patients
Acronym: IHDIP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Formación e Investigación de los Profesionales de la Salud de Extremadura (Other)
Collaborators: Hospital Arquitecto Marcide. Ferrol. A Coruña. (Spain) (Unknown); Hospital San Pedro de Alcantara (Other); Virgen del Puerto Hospital (Other); Hospital Central de la Defensa Gómez Ulla. Madrid (Spain) (Unknown); Hospital Costa del Sol (Other); Hospital Obispo Polanco. Teruel (Spain) (Unknown); Hospital de Manises. Valencia (Spain) (Unknown); Hospital Virgen de la Concha. Zamora (Spain) (Unknown); Hospital de Especialidades de las Fuerzas Armadas. Quito (Ecuador) (Unknown); Servicio Extremeño de Salud (Spain) (Unknown); Hospital del SAS de Jerez (Other); Hospital Nuestra Sra de Sonsoles. Ávila (Spain) (Unknown); Dialysis Center SM2. Potenza (Italy) (Unknown); Miulli General Hospital (Other); Hospital del Rio Hortega (Other); Hospital Duran de Buenos Aires (Unknown); Hospital El Bierzo (Other); Hospitales Universitarios Virgen del Rocío (Other); Hospital Universitario Virgen Macarena (Other); University Hospital of Girona Dr. Josep Trueta (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IHDIP (P1712)
Record Dates: First submitted 2017-07-04; First posted 2017-08-04 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Renal Disease, End-Stage
Keywords: once-weekly haemodialysis; incremental haemodialysis; randomized clinical trial
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicenter, randomized clinical trial. It has two strata: for age (≥or< 75 years old) and for KrU (≥or< 5,5 ml/min/1.73m2). It is controlled through usual clinical practice.
  Intervention consists in reducing the frequency or number of sessions per week with which patients start the HD treatment. The experimental group will start with one session/week, then the number of weekly sessions will be increased to two and later to three as per criteria for progression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 76 patients who start RRT with the incremental HD regimen.
  Interventions: Procedure: Incremental haemodialysis
- Control group (Active Comparator): 76 patients who start RRT with the conventional HD (3 sessions per week)
  Interventions: Procedure: Conventional haemodialysis

INTERVENTIONS:
Procedure: Incremental haemodialysis — It consists in reducing the frequency or number of sessions per week with which patients start the HD treatment. The experimental group will start with one session/week, then the number of weekly sessions will be increased to two and later to three as per criteria for progression
  Arms: Experimental group
Procedure: Conventional haemodialysis — It is controlled through usual clinical practice, based on starting the HD treatment with three sessions per week (control group).
  Arms: Control group

SUMMARY:
Background: Incremental hemodialysis (HD) is a starting regime for renal replacement therapy (RRT) adapted to each patient's necessities. It is mainly conditioned by the residual renal function (RRF). The frequency of sessions with which patients start HD -one or two sessions per week-, is lower than that for conventional HD three times per week. Such frequency is increased (from one to two sessions, and from two to three sessions) as the RRF declines.

Methods/Design: IHDIP is a multicenter randomized experimental open trial. It is randomized in a 1:1 ratio and controlled through usual clinical practice, with a low intervention level and non-commercial. It includes 152 patients older than 18 years with chronic renal disease stage 5 and start HD as RRT, with a RRF of ≥ 4ml/min/1.73m2, measured by renal clearance of urea (KrU). The intervention group includes 76 patients who will start with one session of HD per week (incremental HD). The control group includes 76 patients who will start with three sessions per week (conventional HD). The primary purpose is assessing the survival rate, while the secondary purposes are the morbidity rate (hospital admissions), the clinical parameters, the quality of life and the efficiency.

Discussion: This study will enable us to know with the highest level of scientific evidence, the number of sessions a patient should receive when starting the HD treatment, depending on his/her RRF.

DETAILED DESCRIPTION:
Conventional thrice-weekly HD for 3 to 5 hours in a health center in an outpatient basis is the most used renal replacement therapy (RRT) regimen (1). However, it has an unacceptable high mortality rate (10%-20% a year). In order to try to improve those results, new regimens have been proposed. They are based on an increase of the HD dose and/or a higher number of sessions (2). Nevertheless, inconsistent results in terms of clinical benefits with such programs have been shown in recently published randomized and controlled trials (3,4), together with a lower rate of vascular access success (5) and a lower maintenance of the RRF (6) The National Kidney Foundation-Kidney Disease Outcomes Quality Initiate (NKD KDOQI 2015)(1) 2015 guidelines allow the reduction in the weekly HD dose for patients with a residual kidney urea clearance (KrU) higher than 3ml/min/1.73m2. In these cases, the renal clearance (Kr) is added to the dialysis clearance (Kd) obtained in 2 sessions per week, thus obtaining the adequate dialysis dose (7,8) Surprisingly enough, few centers follow this recommendation when over 50% of patients start HD with KrU >3 mL/min (9).

Authors like Kalantar-Zadeh et al (9,10) in the U.S.A. or Teruel et al (11) in Spain have published their experience with 2 HD sessions per week in incident patients. Through this regime they have shown that the RRF is preserved and the survival rate is similar to the one obtained with the conventional HD. This is due to the fact that the Kr has much greater clinical weight than Kd7, since the RRF contributes to the production of vitamin D and erythropoietine (12,13), and eliminates the protein-bound uremic toxins that are poorly dialyzed (13,14). In other words, the RRF plays a fundamental role both in the dialysis adequacy and in survival (15,16).

Currently, some authors are questioning the number of HD sessions with which a patient should start the renal replacement therapy (RRT) (7, 17-19). Progressive HD is an initiation regimen adapted to the patient's RRF. The frequency increases as the daily diuretic level declines (7, 17-19).

The IHDIP trial20 aims at determining whether or not starting with one HD session per week reduces mortality in incident patients and its influence in morbidity (hospital admissions), clinical parameters, quality of life and efficiency with regard to the patients who start RRT with the conventional method.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged >18 years, incident patients with stage 5 CKD who have chosen HD as RRT initiation.
* RRF measured by KrU ≥ 4 ml/min/1.73m2. In general, it is advised not to start HD with a KrU> 7.
* Informed consent signed before starting any activity related to the trial.

Exclusion Criteria:

* Unplanned HD initiation (established in point 7.4 of the protocol)
* Non incident patients, in other words, patients who were previously on RRT, either on peritoneal dialysis, or on kidney transplant.
* Active neoplasia at the moment of inclusion
* Cardiovascular disease defined as: heart failure type IV of the New York Heart Association (NYHA), unstable angina or ischemic cardiopathy which has caused any admission in hospital in the last 3 months.
* Cardiorenal syndrome
* Active inflammatory disease with immunosuppressive treatment
* Hepatorenal syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 24 months
  Assess and compare survival in subjects with one session a week as an RRT starting regimen, compared to those patients who start RRT with the conventional method

SECONDARY OUTCOMES:
Hospital admissions | 24 months
  Number of hospitalizations, for any cause; and number of days hospitalized for any cause
Residual Kidney Function (RRF) maintenance . | 24 months
  Reduction of glomerular filtration rate (GFR) and tubular function. Average urine volume and percentage of patients with anuria (≤200ml/day in two consecutive measurements).
Analysis of anemia | 3, 6, 9, 12, 18 and 24 months
  Mean hemoglobin levels and Proportion of patients with Hb measurement inside the target range (10.5-12 g/dl) and The erythropoietin resistance index (ERI): ERI = weekly EPO (in UI)/patient's weight (in kg)/Hb (in gr/dl)
Bone-mineral metabolism | 3, 6, 9, 12, 18 and 24 months
  Mean levels of calcium, phosphorus and intac PTH levels. Estimate the percentage of patients within the therapeutic range; Calcium 8,4-9,5mg/dl, Phosphorus 3,5-5,5mg/dl and iPTH 150-300 pg/dl.
Hypertrophic cardiomyopathy levels | Basal, anual and end of the follow-un visit
Estimation of the effect of treatment on quality of life | 3, 6, 9, 12, 18 and 24 months
  Quality of life survey values from Kidney Disease and Quality of Life (KDQOL'36 Spanish) will be registered.
Assessing RRT efficiency (costs) | 12 and 24 months
  The number of sessions perform in subjects of incremental HDF group Vs number of sessions in the conventional HD group. The cost of each session is defined by the public contest for private haemodialysis clinics arranged by (that work to) the Health Service of Extremadura.

CONTACTS AND LOCATIONS:
Overall Officials: Javier L Deira Lorenzo, PhD MD, Principal Investigator — Servicio Extremeño de Salud; Miguel A Suarez Santisteban, MD, Principal Investigator — Servicio Extremeño de Salud
Locations (3):
- Spain (3):
  - FundeSalud. Junta de Extremadura, Mérida, Badajoz
  - Hospital Virgen del Puerto, Plasencia, Cáceres
  - Hospital San Pedro de Alcántara, Cáceres

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] National Kidney Foundation. KDOQI Clinical Practice Guideline for Hemodialysis Adequacy: 2015 update. Am J Kidney Dis. 2015 Nov;66(5):884-930. doi: 10.1053/j.ajkd.2015.07.015. PMID 26498416
- [Background] Chan CT, Covic A, Craig JC, Davenport A, Kasiske BL, Kuhlmann MK, Levin NW, Li PK, Locatelli F, Rocco MV, Wheeler DC. Novel techniques and innovation in blood purification: a clinical update from Kidney Disease: Improving Global Outcomes. Kidney Int. 2013 Mar;83(3):359-71. doi: 10.1038/ki.2012.450. Epub 2013 Jan 16. PMID 23325091
- [Background] Chertow GM, Levin NW, Beck GJ, Daugirdas JT, Eggers PW, Kliger AS, Larive B, Rocco MV, Greene T; Frequent Hemodialysis Network (FHN) Trials Group. Long-Term Effects of Frequent In-Center Hemodialysis. J Am Soc Nephrol. 2016 Jun;27(6):1830-6. doi: 10.1681/ASN.2015040426. Epub 2015 Oct 14. PMID 26467779
- [Background] Rocco MV, Daugirdas JT, Greene T, Lockridge RS, Chan C, Pierratos A, Lindsay R, Larive B, Chertow GM, Beck GJ, Eggers PW, Kliger AS; FHN Trial Group. Long-term Effects of Frequent Nocturnal Hemodialysis on Mortality: The Frequent Hemodialysis Network (FHN) Nocturnal Trial. Am J Kidney Dis. 2015 Sep;66(3):459-68. doi: 10.1053/j.ajkd.2015.02.331. Epub 2015 Apr 8. PMID 25863828
- [Background] Suri RS, Larive B, Sherer S, Eggers P, Gassman J, James SH, Lindsay RM, Lockridge RS, Ornt DB, Rocco MV, Ting GO, Kliger AS; Frequent Hemodialysis Network Trial Group. Risk of vascular access complications with frequent hemodialysis. J Am Soc Nephrol. 2013 Feb;24(3):498-505. doi: 10.1681/ASN.2012060595. Epub 2013 Feb 7. PMID 23393319
- [Background] Daugirdas JT, Greene T, Rocco MV, Kaysen GA, Depner TA, Levin NW, Chertow GM, Ornt DB, Raimann JG, Larive B, Kliger AS; FHN Trial Group. Effect of frequent hemodialysis on residual kidney function. Kidney Int. 2013 May;83(5):949-58. doi: 10.1038/ki.2012.457. Epub 2013 Jan 23. PMID 23344474
- [Background] Clark EG, Bagshaw SM. Unnecessary renal replacement therapy for acute kidney injury is harmful for renal recovery. Semin Dial. 2015 Jan-Feb;28(1):6-11. doi: 10.1111/sdi.12300. Epub 2014 Oct 30. PMID 25359104
- [Background] Mathew AT, Fishbane S, Obi Y, Kalantar-Zadeh K. Preservation of residual kidney function in hemodialysis patients: reviving an old concept. Kidney Int. 2016 Aug;90(2):262-271. doi: 10.1016/j.kint.2016.02.037. Epub 2016 May 12. PMID 27182000
- [Background] Patel N, Hu SL. Preserving residual renal function in dialysis: what we know. Semin Dial. 2015 May-Jun;28(3):250-8. doi: 10.1111/sdi.12302. Epub 2014 Sep 18. PMID 25231758
- [Background] Casino FG, Basile C. The variable target model: a paradigm shift in the incremental haemodialysis prescription. Nephrol Dial Transplant. 2017 Jan 1;32(1):182-190. doi: 10.1093/ndt/gfw339. PMID 27742823
- [Background] Shafi T, Jaar BG, Plantinga LC, Fink NE, Sadler JH, Parekh RS, Powe NR, Coresh J. Association of residual urine output with mortality, quality of life, and inflammation in incident hemodialysis patients: the Choices for Healthy Outcomes in Caring for End-Stage Renal Disease (CHOICE) Study. Am J Kidney Dis. 2010 Aug;56(2):348-58. doi: 10.1053/j.ajkd.2010.03.020. Epub 2010 Jun 3. PMID 20605303
- [Background] van der Wal WM, Noordzij M, Dekker FW, Boeschoten EW, Krediet RT, Korevaar JC, Geskus RB; Netherlands Cooperative Study on the Adequacy of Dialysis Study Group (NECOSAD). Full loss of residual renal function causes higher mortality in dialysis patients; findings from a marginal structural model. Nephrol Dial Transplant. 2011 Sep;26(9):2978-83. doi: 10.1093/ndt/gfq856. Epub 2011 Feb 11. PMID 21317411
- [Background] Obi Y, Streja E, Rhee CM, Ravel V, Amin AN, Cupisti A, Chen J, Mathew AT, Kovesdy CP, Mehrotra R, Kalantar-Zadeh K. Incremental Hemodialysis, Residual Kidney Function, and Mortality Risk in Incident Dialysis Patients: A Cohort Study. Am J Kidney Dis. 2016 Aug;68(2):256-265. doi: 10.1053/j.ajkd.2016.01.008. Epub 2016 Feb 9. PMID 26867814
- [Background] Wong J, Vilar E, Davenport A, Farrington K. Incremental haemodialysis. Nephrol Dial Transplant. 2015 Oct;30(10):1639-48. doi: 10.1093/ndt/gfv231. Epub 2015 Jun 1. PMID 26038351
- [Background] Termorshuizen F, Dekker FW, van Manen JG, Korevaar JC, Boeschoten EW, Krediet RT; NECOSAD Study Group. Relative contribution of residual renal function and different measures of adequacy to survival in hemodialysis patients: an analysis of the Netherlands Cooperative Study on the Adequacy of Dialysis (NECOSAD)-2. J Am Soc Nephrol. 2004 Apr;15(4):1061-70. doi: 10.1097/01.asn.0000117976.29592.93. PMID 15034110
- [Background] Vilar E, Wellsted D, Chandna SM, Greenwood RN, Farrington K. Residual renal function improves outcome in incremental haemodialysis despite reduced dialysis dose. Nephrol Dial Transplant. 2009 Aug;24(8):2502-10. doi: 10.1093/ndt/gfp071. Epub 2009 Feb 24. PMID 19240122
- [Background] Zhang M, Wang M, Li H, Yu P, Yuan L, Hao C, Chen J, Kalantar-Zadeh K. Association of initial twice-weekly hemodialysis treatment with preservation of residual kidney function in ESRD patients. Am J Nephrol. 2014;40(2):140-50. doi: 10.1159/000365819. Epub 2014 Aug 23. PMID 25171342
- [Background] Fernandez Lucas M, Teruel JL. Incremental hemodialysis schedule at the start of renal replacement therapy. Nefrologia. 2017 Jan-Feb;37(1):1-4. doi: 10.1016/j.nefro.2016.08.002. Epub 2016 Oct 1. No abstract available. English, Spanish. PMID 27707578
- [Background] Toth-Manikowski SM, Shafi T. Hemodialysis Prescription for Incident Patients: Twice Seems Nice, But Is It Incremental? Am J Kidney Dis. 2016 Aug;68(2):180-183. doi: 10.1053/j.ajkd.2016.04.005. No abstract available. PMID 27477358
- [Background] Caria S, Cupisti A, Sau G, Bolasco P. The incremental treatment of ESRD: a low-protein diet combined with weekly hemodialysis may be beneficial for selected patients. BMC Nephrol. 2014 Oct 29;15:172. doi: 10.1186/1471-2369-15-172. PMID 25352299
- [Background] Bolasco P, Cupisti A, Locatelli F, Caria S, Kalantar-Zadeh K. Dietary Management of Incremental Transition to Dialysis Therapy: Once-Weekly Hemodialysis Combined With Low-Protein Diet. J Ren Nutr. 2016 Nov;26(6):352-359. doi: 10.1053/j.jrn.2016.01.015. Epub 2016 Feb 28. PMID 26936151
- [Background] Libetta C, Esposito P, Dal Canton A. Once-weekly hemodialysis: a single-center experience. Am J Kidney Dis. 2015 Feb;65(2):343. doi: 10.1053/j.ajkd.2014.07.034. No abstract available. PMID 25616635
- [Background] Parra Moncasi E, Arenas Jimenez MD, Alonso M, Martinez MF, Gamen Pardo A, Rebollo P, Ortega Montoliu T, Martinez Terrer T, Alvarez-Ude F; Grupo de Gestion de la Calidad de la Sociedad Espanola de Nefrologia. Multicentre study of haemodialysis costs. Nefrologia. 2011;31(3):299-307. doi: 10.3265/Nefrologia.pre2011.Apr.10813. English, Spanish. PMID 21629336
- [Derived] Deira J, Suarez MA, Lopez F, Garcia-Cabrera E, Gascon A, Torregrosa E, Garcia GE, Huertas J, de la Flor JC, Puello S, Gomez-Raja J, Grande J, Lerma JL, Corradino C, Musso C, Ramos M, Martin J, Basile C, Casino FG. IHDIP: a controlled randomized trial to assess the security and effectiveness of the incremental hemodialysis in incident patients. BMC Nephrol. 2019 Jan 9;20(1):8. doi: 10.1186/s12882-018-1189-6. PMID 30626347
- [Derived] Suarez MA, Garcia-Cabrera E, Gascon A, Lopez F, Torregrosa E, Garcia GE, Huertas J, de la Flor JC, Puello S, Gomez-Raja J, Grande J, Lerma JL, Corradino C, Ramos M, Martin J, Basile C, Casino FG, Deira J. Rationale and design of DiPPI: A randomized controlled trial to evaluate the safety and effectiveness of progressive hemodialysis in incident patients. Nefrologia (Engl Ed). 2018 Nov-Dec;38(6):630-638. doi: 10.1016/j.nefro.2018.07.010. Epub 2018 Oct 19. English, Spanish. PMID 30344012

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT03239808/Prot_SAP_000.pdf
  • Informed Consent Form (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT03239808/ICF_001.pdf